CLINICAL TRIAL: NCT01628874
Title: A Double-Blind, Randomized Controlled Trial of Jet Injection of 1% Buffered Lidocaine Versus Topical EMLA for Local Anesthesia Before Lumbar Puncture in Children
Brief Title: Jet Injection of 1% Buffered Lidocaine Versus Topical EMLA for Local Anesthesia Before Lumbar Puncture in Children
Acronym: JTIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low recruitment numbers, the study was terminated.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-0542
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Lumbar Puncture; Topical Analgesia
Keywords: Lumbar Puncture; J-Tip; Jet injection; Local Analgesia
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine Injection (Experimental): 0.5 mL (5mg) of 1% lidocaine injection given with the J-Tip
  Interventions: Device: J-Tip; Drug: EMLA; Drug: Lidocaine
- lidocaine 2.5% and prilocaine 2.5% (EMLA) Cream (Active Comparator): Patients in this arm will receive 1g EMLA cream if they are in the younger age group and 10g EMLA cream if they are in the older age group. This will be placed for a minimum of 30 minutes.
  Interventions: Device: J-Tip; Drug: EMLA; Drug: Lidocaine

INTERVENTIONS:
Device: J-Tip — Used once for both arms prior to lumbar puncture. The Experimental arm will receive 0.5 mL (5mg) of 1% Lidocaine. The Active Comparator arm will receive normal saline. This will occur after the cream has been placed for 30 minutes and wiped away and prior to the lumbar puncture.
  Other Names: Needle-free jet-injection system
Drug: EMLA — In the Active Comparator arm, lidocaine 2.5% and prilocaine 2.5% cream placed over area where lumbar puncture will occur for at least 30 minutes. This same procedure will occur for the Experimental arm with a placebo cream instead. This will occur once prior to the J-Tip injection and lumbar puncture.
  Other Names: EMLA Cream
Drug: Lidocaine — 5 mg given via J-Tip once, repeat dosing as needed in the Experimental group. A placebo will be given in the Active Comparator group.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a needle-free jet-injection system with 1% buffered lidocaine for local anesthesia for lumbar punctures compared to a topical anesthetic agent. Our hypothesis is: A needle-free jet-injection system (J-Tip) with 1% lidocaine will provide local anesthesia that is comparable to that of a topical anesthetic agent (EMLA cream) when performing lumbar punctures in children.

DETAILED DESCRIPTION:
Lumbar punctures are a common procedure performed in children in the emergency department. In febrile infants they are frequently performed as part of a sepsis evaluation, and in older children they are used in the evaluation of possible meningitis, new seizures, altered mental status and other neurologic emergencies.

Several studies in the pediatric emergency medicine literature have found a positive association between lumbar puncture success and the use of local anesthesia in infant lumbar punctures. Despite this data, studies have shown that 70-76% of lumbar punctures in the emergency department are performed without any form of pain management, with up to 95% of infants receiving no form of pain management. Common reasoning for providers to forgo pain management include the time for topical anesthetics to be effective (30-45 minutes), the pain already associated with injectable lidocaine, and obscuring of anatomic landmarks with injectable lidocaine.

A recent development in pain management for pediatric procedures is the use of needle-free jet injection of lidocaine. One such device is the J-Tip, which uses a compressed carbon dioxide (CO2) cartridge to deliver medication to the subcutaneous tissues to a depth of 5-8 mm in 0.2 seconds. It has been shown to be largely pain-free for children. Multiple studies have shown it to be effective in reducing pain associated with peripheral IV placement in children. The J-Tip has recently been approved for peripheral IV starts in the Children's Hospital Colorado emergency department.

Some hospitals anecdotally report using the device for lumbar punctures, but to date no randomized studies have evaluated its effectiveness in pain management compared to other methods. Our study aims to evaluate the efficacy of the J-Tip in lumbar punctures. It offers the advantage of providing much faster anesthesia compared to topical creams, yet does not require the initial skin puncture of injectable lidocaine. If a rapid form of local anesthesia is available, it may increase the overall use of local anesthesia and improve pain management in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* age ≤4 months or 4-18 years
* ability to report VAS for patients 4-18 years
* require lumbar puncture as part of their clinical care

Exclusion Criteria:

* ages 5-47 months
* developmental delay or inability to complete VAS in older patients
* allergy to lidocaine
* requirement of sedation for procedure
* pre-procedural analgesia treatment except for nonsteroidal anti-inflammatory drugs and acetaminophen.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2012-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Caltagirone, MD, Principal Investigator — Children's Hospital Colorado and University of Colorado Denver; Kathleen Adelgais, MD, MPH, Principal Investigator — Children's Hospital Colorado and University of Colorado Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Background] Fein D, Avner JR, Khine H. Pattern of pain management during lumbar puncture in children. Pediatr Emerg Care. 2010 May;26(5):357-60. doi: 10.1097/PEC.0b013e3181db2026. PMID 20404782
- [Background] Baxter AL, Welch JC, Burke BL, Isaacman DJ. Pain, position, and stylet styles: infant lumbar puncture practices of pediatric emergency attending physicians. Pediatr Emerg Care. 2004 Dec;20(12):816-20. doi: 10.1097/01.pec.0000148030.99339.fe. PMID 15572969
- [Background] Spanos S, Booth R, Koenig H, Sikes K, Gracely E, Kim IK. Jet Injection of 1% buffered lidocaine versus topical ELA-Max for anesthesia before peripheral intravenous catheterization in children: a randomized controlled trial. Pediatr Emerg Care. 2008 Aug;24(8):511-5. doi: 10.1097/PEC.0b013e31816a8d5b. PMID 18645542
- [Background] Quinn M, Carraccio C, Sacchetti A. Pain, punctures, and pediatricians. Pediatr Emerg Care. 1993 Feb;9(1):12-4. doi: 10.1097/00006565-199302000-00005. No abstract available. PMID 8488137
- [Background] Tomlinson D, von Baeyer CL, Stinson JN, Sung L. A systematic review of faces scales for the self-report of pain intensity in children. Pediatrics. 2010 Nov;126(5):e1168-98. doi: 10.1542/peds.2010-1609. Epub 2010 Oct 4. PMID 20921070
- [Background] Baxter AL, Fisher RG, Burke BL, Goldblatt SS, Isaacman DJ, Lawson ML. Local anesthetic and stylet styles: factors associated with resident lumbar puncture success. Pediatrics. 2006 Mar;117(3):876-81. doi: 10.1542/peds.2005-0519. PMID 16510670
- [Background] Powell CV, Kelly AM, Williams A. Determining the minimum clinically significant difference in visual analog pain score for children. Ann Emerg Med. 2001 Jan;37(1):28-31. doi: 10.1067/mem.2001.111517. PMID 11145767
- [Background] Nigrovic LE, Kuppermann N, Neuman MI. Risk factors for traumatic or unsuccessful lumbar punctures in children. Ann Emerg Med. 2007 Jun;49(6):762-71. doi: 10.1016/j.annemergmed.2006.10.018. Epub 2007 Feb 23. PMID 17321005
- [Background] Jimenez N, Bradford H, Seidel KD, Sousa M, Lynn AM. A comparison of a needle-free injection system for local anesthesia versus EMLA for intravenous catheter insertion in the pediatric patient. Anesth Analg. 2006 Feb;102(2):411-4. doi: 10.1213/01.ane.0000194293.10549.62. PMID 16428534
- [Background] Kaur G, Gupta P, Kumar A. A randomized trial of eutectic mixture of local anesthetics during lumbar puncture in newborns. Arch Pediatr Adolesc Med. 2003 Nov;157(11):1065-70. doi: 10.1001/archpedi.157.11.1065. PMID 14609894
- [Background] Rushforth JA, Levene MI. Behavioural response to pain in healthy neonates. Arch Dis Child Fetal Neonatal Ed. 1994 May;70(3):F174-6. doi: 10.1136/fn.70.3.f174. PMID 8198409
- [Background] Grunau RVE, Craig KD. Pain expression in neonates: facial action and cry. Pain. 1987 Mar;28(3):395-410. doi: 10.1016/0304-3959(87)90073-X. PMID 3574966
- [Derived] Caltagirone R, Raghavan VR, Adelgais K, Roosevelt GE. A Randomized Double Blind Trial of Needle-free Injected Lidocaine Versus Topical Anesthesia for Infant Lumbar Puncture. Acad Emerg Med. 2018 Mar;25(3):310-316. doi: 10.1111/acem.13351. Epub 2017 Dec 26. PMID 29160002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to low enrollment, the study was halted prior to getting to the planned protocol enrollment. The patients who were enrolled were used in the analysis per the participant flow module.
Groups:
- EMLA Cream, Then Placebo Via J-Tip: Patients in this arm received 1g EMLA cream (lidocaine 2.5% and prilocaine 2.5%) placed on the lumbar puncture site for a minimum of 30 minutes. The cream was then wiped away, and they were given 0.5 mL NS placebo injection via the J-Tip at the lumbar puncture site.
- Placebo Cream, Then Lidocaine Via J-Tip: Participants in this arm had placebo cream placed on the lumbar puncture site for minimum of 30 minutes. The cream was then wiped away, and they were given 0.5 mL (5mg) of 1% lidocaine injection via the J-Tip at the lumbar puncture site.
Period: Overall Study
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip
Started | 34 | 32
Completed | 29 | 29
Not Completed | 5 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Age >4 months | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 30 [19 to 48] | 41 [28 to 50] | 35.5 [20 to 51.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 7 | 8
  White | 20 | 16 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: The pain score was assessed using the 5-point Neonatal Coding System (NFCS) on a scale of 0-5, with 0 indicating no pain and 5 the highest level of pain.
Time Frame: Immediately Post-Procedure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip
Number analyzed (Participants) | 29 | 29
score on a scale | 0 [0 to 0.5] | 0 [0 to 0]

2. Primary Outcome: Pain Score
Description: as for outcome 1
Time Frame: At Needle Insertion
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip
Number analyzed (Participants) | 29 | 29
score on a scale | 5 [5 to 5] | 5 [4 to 5]

3. Primary Outcome: Pain Score
Description: as for outcome 1
Time Frame: At time J-TIP is used
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip
Number analyzed (Participants) | 29 | 29
score on a scale | 5 [5 to 5] | 5 [5 to 5]

4. Secondary Outcome: Number of Participants With Lumbar Puncture Success
Description: The success of lumbar puncture was defined as obtaining Cerebrospinal fluid (CSF) on the first attempt and <1000 Red Blood Cells/millimeter cubed
Time Frame: Immediately following lumbar puncture
Measure: Count of Participants; unit: Participants
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip
Number analyzed (Participants) | 29 | 29
Participants | 8 | 16

5. Secondary Outcome: Change in Heart Rate
Description: Heart rate was measured at 5 points in time (pre-procedure, application of J-Tip, at LP needle insertion, while the needle is in place, and post-procedure) and was compared for significant differences
Time Frame: At 5 specific points during the procedure
Measure: Mean (Standard Deviation); unit: Beats per Minute
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip
Number analyzed (Participants) | 29 | 29
Beats per Minute
  Pre-procedure | 154 (40) | 156 (28)
  J-Tip application | 160 (37) | 167 (29)
  Needle insertion | 170 (49) | 169 (35)
  Needle in place | 172 (54) | 178 (40)
  Post-procedure | 157 (30) | 159 (26)

ADVERSE EVENTS:
Arm/Group | EMLA Cream, Then Placebo Via J-Tip | Placebo Cream, Then Lidocaine Via J-Tip
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 0/34 | 0/32

LIMITATIONS AND CAVEATS:
Low enrollment leading to small number of subjects analyzed; Low enrollment of older age range (4 years-18 years) leading to termination of that study arm prior to analysis (6 subjects excluded from analysis, no data for VAS collected).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No